CLINICAL TRIAL: NCT01311349
Title: Evaluation of the Antimicrobial Activity In Vitro of Tigecycline in Comparison to Other Broad Spectrum Antibiotics in Isolates Collected From Patients
Brief Title: Study Evaluating Local Susceptibility Patterns Associated With Tigecycline in Comparison to Other Antibiotics
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 3074A1-102056
Record Dates: First submitted 2009-08-10; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2009-08

CONDITIONS: Infection
Keywords: Susceptibility of tigecycline; Drug Resistance, Bacterial
MeSH Terms: conditions — Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: A listing of all isolates meeting the inclusion criteria will be maintained.

SUMMARY:
Various bacterial organisms will be tested in order to compile information regarding the effectiveness of tigecycline against certain bacteria seen in local communities.

DETAILED DESCRIPTION:
This is a prospective, microbiologic in vitro evaluation which will study the susceptibility of tigecycline in disk diffusion on clinical bacterial isolates collected from inpatients and outpatients. Fourteen hospital centers participated in the program. In vitro efficacy of tigecycline will be determined through the in vitro disk diffusion activity, using FDA breakpoints.

ELIGIBILITY:
Inclusion Criteria: Any protocol-specified microorganism isolated from the samples collected from hospitalized patients and outpatients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients and outpatients
Sampling Method: Probability Sample
Enrollment: 1575 (Actual)
Dates: Start 2005-12; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer